CLINICAL TRIAL: NCT02043171
Title: Year-long Double Blind Study on the Efficacy of a Combination of Beta-hydroxy-beta-methylbutyrate and Vitamin D With and Without Exercise on Muscular Strength and Functionality in Older Adults.
Brief Title: Nutritional Intervention for Age-related Muscular Function and Strength Losses-Study 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: Iowa State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTI2014-CS01
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Vitamin D; Cholecalciferol; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo Exercise (Placebo Comparator): Placebo supplementation group with 3 days per week of exercise
  Interventions: Dietary Supplement: Placebo; Behavioral: Exercise
- Placebo Non-exercise (Placebo Comparator): Placebo supplementation group without exercise
  Interventions: Dietary Supplement: Placebo; Behavioral: Non-Exercise
- HMB plus Vitamin D Exercise (Active Comparator): HMB plus Vitamin D supplementation group with 3 days per week of exercise
  Interventions: Drug: HMB plus Vitamin D; Behavioral: Exercise
- HMB plus Vitamin D Non-exercise (Active Comparator): HMB plus Vitamin D supplementation group without exercise
  Interventions: Drug: HMB plus Vitamin D; Behavioral: Non-Exercise

INTERVENTIONS:
Dietary Supplement: Placebo — A Placebo comparator
  Arms: Placebo Exercise; Placebo Non-exercise
Drug: HMB plus Vitamin D — Active comparator of HMB (3 g/d) plus Vitamin D (2,000 IU/d)
  Other Names: HMB (Calcium beta-hydroxy-beta-methylbutyrate); Vitamin D (Cholecalciferol)
  Arms: HMB plus Vitamin D Exercise; HMB plus Vitamin D Non-exercise
Behavioral: Non-Exercise — This group will not participate in 3 times per week strength training
  Arms: HMB plus Vitamin D Non-exercise; Placebo Non-exercise
Behavioral: Exercise — This group will participate in a supervised 3 times per week strength training program
  Arms: HMB plus Vitamin D Exercise; Placebo Exercise

SUMMARY:
Men and women lose muscle mass and strength with age. Loss of muscle mass and strength is accompanied by a loss of muscle function which can lead to diminished quality of life and more importantly can lead to serious fall requiring medical treatment. The investigators hypothesize that the combined supplements of Calcium-HMB and Vitamin D will lead to decreased falls and to improved quality of life (QOL) for older adults. The investigators further hypothesize that the addition of a modest exercise regimen to these supplements will enhance the synergistic effects of both Calcium-HMB and Vitamin D.

Subjects will consume the dietary supplement 2 times per day for 12 months. Tests will consist of the following: a) strength of subjects' legs and elbow by Isokinetic Dynamometer; b) body composition; c) hand-grip strength by hand-grip dynamometer; d) functional mobility, balance and agility (Get-Up and Get-Up-and-Go tests); e) filling out questionnaires; and g) having blood drawn for biochemical measurements. Testing will be performed at the baseline (0 months) and at 3, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects will be enrolled into the study.
* Age > 60 years.
* Free of liver and kidney diseases, and with no evidence of uncontrolled hypertension.
* Does not have a chronic disease that affects calcium or bone metabolism (i.e., asthma with chronic use of high dose steroids, inflammatory bowel disease, Crohn's disease, primary hyperparathyroidism, seizure disorder with use of phenobarbital, etc.).
* Not classified as morbidly obese (body mass index (BMI) >40 kg/m2).
* Six weeks since major surgery (three weeks since minor surgery).
* Willing to consume one of the nutritional supplements for the study period.
* Individuals diagnosed with osteoporosis, or bone density > 2.0 standard deviations below the mean, will not be enrolled in the study.
* No other serious medical illness.
* Serum 25OH-vitD3 >15 ng/ml.
* Willing to participate in 3-day-a-week monitored strength-training program.
* Physician has placed no restriction on physical exercise.

Exclusion Criteria:

* Age < 60 years.
* Evidence of liver and kidney diseases, uncontrolled hypertension, or Type I diabetes mellitus requiring insulin for glucose control.
* Presence of a chronic disease that affects calcium or bone metabolism (i.e., asthma with chronic use of high dose steroids, inflammatory bowel disease, Crohn's disease, primary hyperparathyroidism, seizure disorder with use of phenobarbital, etc.).
* Classified as morbidly obese (body mass index (BMI) >40 kg/m2).
* Less than six weeks since major surgery or three weeks since minor surgery.
* Not willing to consume one of the nutritional supplements for the study period.
* Individuals diagnosed with osteoporosis, or a bone density > 2.0 standard deviations below the mean, will not be enrolled in the study.
* Other serious medical illness, which the subject's doctor or medical review team has decided affects the subject's ability to participate in the study.
* History of blood clots and/or the use of blood thinning medications
* Subjects on high dose vitamin D therapies (i.e. 50,000 IU vitamin D).
* Subjects with serum 25OH-vitD3 <10 ng/ml will be considered deficient and will be referred to their physician for treatment.
* Subjects with serum 25OH-vitD3 >30 ng/ml may not respond to the intervention as expected and will also be excluded from the study.
* Not able or willing to participate in 3-day-a-week monitored strength-training program.
* Physician has placed a restriction on physical exercise.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Muscular strength | 12 Months
  Leg and elbow strength will be tested by Isokinetic dynamometer and Handgrip strength will be tested using a hand-grip dynamometer.

SECONDARY OUTCOMES:
Functionality | 12 months
  The Get-Up and Get-Up-and-Go tests will be used as a measure of functionality.

OTHER OUTCOMES:
Muscle mass | 12 months
  Body composition will be measured by bioelectrical impedance analysis (BIA)and dual-energy X-ray absorptiometry (DXA), and air displacement plethysmography (BODPOD) during the study.
Quality of life | 12 months
  Questionnaires will be administered to assess feeling, general health, the IPAQ, cognitive functioning, and SF-36.

CONTACTS AND LOCATIONS:
Overall Officials: John A Rathmacher, PhD, Principal Investigator — Metabolic Technologies Inc.
Locations (1):
- Iowa State University, Ames, Iowa, United States